CLINICAL TRIAL: NCT00981097
Title: Evaluation of Serum Free Light Chains and Clonal Ig DNA in Plasma From Patients With Aggressive B-Cell Lymphomas
Brief Title: Study of Blood and Tissue Samples From Patients With Aggressive Non-Hodgkin B-Cell Lymphoma or Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMC-064; U01CA121947 (NIH); CDR0000648183 (Other: NCI)
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma; Nonneoplastic Condition
Keywords: HIV infection; HIV-associated Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; HIV Infections; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 tubes of peripheral blood collected along with available tissue blocks or fresh frozen tissue collected at baseline.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimen Collection: Subjects with a diagnosis of HIV and an untreated aggressive B-cell lymphoma.
  Interventions: Genetic: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: polymerase chain reaction — determination of elevated serum FLC and clonal Ig detection rates in plasma and tumor
Other: laboratory biomarker analysis — determination of elevated serum FLC and clonal Ig detection rates in plasma and tumor

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood and tissue samples from patients with aggressive non-Hodgkin B-cell lymphoma or Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the proportion of patients with diffuse large B-cell/immunoblastic and Burkitt histologies with elevated serum free light chains (FLC).
* To estimate the proportion of patients with Hodgkin lymphoma with clonal immunoglobulin (Ig) DNA detection in the plasma.

Secondary

* To estimate the agreement between the detection of a monoclonal Ig DNA spike in plasma and the detection of a monoclonal DNA spike in tumor tissue.
* To estimate the agreement between the fragment length of a spike in tumor tissue and the fragment length of the spike in plasma.
* To estimate the detection rate of elevated FLC in each histology, including diffuse large B-cell/immunoblastic and Burkitt lymphoma.
* To estimate the detection rate of clonal Ig DNA in each histology, including diffuse large B-cell/immunoblastic, Burkitt lymphoma, and Hodgkin lymphoma.
* To analyze clinical and pathologic correlates of detection by the serum/plasma tests: disease subtype, stage of disease, disease bulk, lactate dehydrogenase, and Ki-67 index.
* To estimate the detection rate of clonotypic B-cells in peripheral blood mononuclear cells from patients with Hodgkin lymphoma.

OUTLINE: This is a multicenter study.

Blood and tissue samples collected at the time of diagnosis are analyzed for serum free light chain and clonal immunoglobulin (Ig) DNA rearrangements and circulating clonotypic B-cells via PCR.

PROJECTED ACCRUAL: A total of 50 patients (25 with diffuse large B-cell/immunoblastic histologies, 15 with Burkitt lymphoma, and 10 with Hodgkin lymphoma) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of an untreated aggressive B-cell lymphoma, including:

  * Diffuse large B cell/immunoblastic lymphoma
  * Burkitt lymphoma
  * Hodgkin lymphoma
* Serological documentation of HIV infection by any of the FDA-approved tests
* Available diagnostic material from fresh frozen tissue or formalin-fixed paraffin embedded tissue OR willing to undergo a repeat biopsy (fine needle aspiration is acceptable)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with HIV infection and a diagnosis of an untreated aggressive B-cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with diffuse large B-cell/immunoblastic and Burkitt histologies with elevated serum free light chains (FLC) | Study entry
Proportion of patients with Hodgkin lymphoma clonal immunoglobulin (Ig) DNA detection in the plasma | Study entry

SECONDARY OUTCOMES:
Agreement between the detection of a monoclonal Ig DNA spike in plasma and the detection of a monoclonal DNA spike in tumor tissue | Study entry
Agreement between the fragment length of a spike in tumor tissue and the fragment length of the spike in plasma | Study entry
Detection rate of elevated FLC in each histology, including diffuse large B-cell/immunoblastic and Burkitt lymphoma | Study entry
Detection rate of clonal Ig DNA in each histology, including diffuse large B-cell/immunoblastic, Burkitt lymphoma, and Hodgkin lymphoma | Study entry
Analysis of the clinical and pathologic correlates of detection by the serum/plasma tests: disease subtype, stage of disease, disease bulk, lactate dehydrogenase, and Ki67 index | Study entry
Detection rate of clonotypic B cells in peripheral blood mononuclear cells from patients with Hodgkin lymphoma | Study entry

CONTACTS AND LOCATIONS:
Overall Officials: Nina Wagner-Johnston, MD, Principal Investigator — Mallinckrodt Institute of Radiology at Washington University Medical Center
Locations (16):
- United States (16):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - University of California at Davis Center for Aids Research and Education Services, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Mallinckrodt Institute of Radiology at Washington University Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Pennsylvania Oncology Hematology Associates, Incorporated - Philadelphia, Philadelphia, Pennsylvania
  - Thomas Street Health Center, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Wagner-Johnston ND, Lensing S, Noy A, Ratner L, Henry D, Lee JY, Silver S, Faham M, Ambinder RF. High frequency of identical clonal immunoglobulin DNA in pre-treatment tumor and plasma from untreated patients with HIV-associated lymphoma: prospective multicenter trial of the AIDS malignancies consortium (AMC 064). Leuk Lymphoma. 2017 Dec;58(12):2939-2942. doi: 10.1080/10428194.2017.1317095. Epub 2017 May 16. PMID 28508728